CLINICAL TRIAL: NCT06791408
Title: Clinical Study on the Accuracy of Real-time AI-assisted Endocytoscopy in the Diagnosis of Colorectal Diminutive Polyps
Status: Recruiting | Type: Observational
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: 25K014-001
Record Dates: First submitted 2025-01-20; First posted 2025-01-24 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-01

CONDITIONS: Colorectal Polyp

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Colorectal cancer (CRC) is the third most common malignant tumor in the world and the second largest cause of cancer-related death [1]. Colonoscopy is considered the preferred method of screening for colorectal cancer, and early and resectable detection of colorectal neoplastic lesions can significantly reduce colorectal cancer morbidity and mortality. In recent years, with the continuous development of endoscopic diagnostic techniques and the standardization and strengthening of endoscopist training, the detection rate of colorectal polyps has increased year by year. As the number of endoscopic excisions increases, the costs associated with endoscopic excision and pathological diagnosis of excised specimens increase year by year. Research results showed that about 90% of the detected polyps were small polyps (6-9 mm) and diminutive polyps (≤5 mm), and nearly half of them were non-neoplastic polyps, so endoscopic resection and histopathological examination were not required [2, 3]. In order to reduce unnecessary pathological examination and endoscopic treatment, the American Society of Digestive Endoscopy proposed PIVI strategies: "excise and discard" and "diagnose and do not excise" strategies.

Endocytoscopy is a kind of ultra-high magnification endoscopy. Combined with chemical staining and narrow-band imaging technology, endoscopists can observe and judge the nuclear morphology, glandular duct morphology and microvascular morphology of colorectal lesions by naked eye, thus realizing the purpose of real-time biopsy in vivo. However, it takes a lot of experience accumulation to improve the judgment accuracy of endoscopy images, and endoscopy doctors have certain subjective judgments and errors in the process of judging results. Therefore, in order to solve this problem, Artificial Intelligence (AI) is proposed clinically. Our center has developed an artificial intelligence assisted diagnosis system based on endocytoscopy to assist endocytoscopy in judging the nature of colorectal lesions. However, whether this artificial intelligence assisted diagnosis system is accurate in judging the nature of colorectal diminutive polyps and is suitable for widespread promotion and application of PIVI strategy lacks relevant clinical data. This study intends to carry out this clinical study to verify the diagnostic accuracy of this artificial intelligence in the diagnosis of colorectal diminutive polyps.

ELIGIBILITY:
Inclusion Criteria:

* colorectal lesions

Exclusion Criteria:

* lesions lacking high-quality images;
* Inflammatory bowel disease, familial adenomatous polyposis and other special diseases;
* submucosal tumors;
* Pathological diagnosis of inflammatory polyps, Peutz-Jeghers polyps, juvenile polyps, lymphoma and other pathological types.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with colorectal lesions
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Negative predictive value | 2025-12-31
sensitivity | 2025-12-31
specificity | 2025-12-31
accurary | 2025-12-31

CONTACTS AND LOCATIONS:
Overall Officials: Hong Xu, Docror, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China